CLINICAL TRIAL: NCT01707355
Title: Effectiveness of Educational Poster to Primary and Secondary Teachers Regarding Emergency Management of Dental Trauma - A Cluster Randomised Controlled Trial
Brief Title: Effectiveness of Educational Poster to Primary and Secondary Teachers Regarding Emergency Management of Dental Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Cecilia Young, Dr Cecilia Young, The University of Hong Kong
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: HKCTR-1307
Record Dates: First submitted 2012-10-06; First posted 2012-10-16 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Knowledge Regarding Dental Trauma
Keywords: education, knowledge, poster, dental trauma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- invention with poster (Active Comparator): intervention - poster
  Interventions: Behavioral: intervention - poster
- control (No Intervention): control - no poster

INTERVENTIONS:
Behavioral: intervention - poster
  Arms: invention with poster

SUMMARY:
The poster is effective in improving the level of knowledge regarding dental trauma of primary and secondary schools teachers in Hong Kong.

A cluster randomized controlled trial was conducted in mid May 2011,to test the level of knowledge regarding dental trauma with two groups, the intervention group with posters and control group without posters. A questionnaire is used to test the level of knowledge.

DETAILED DESCRIPTION:
A cluster randomized controlled trial was conducted in mid May 2011, Hong Kong where no educational campaign regarding dental trauma targeting on primary and secondary school teachers was implemented before.

Lists of Primary and secondary schools were requested from the Education Bereau. Schools were invited to join the study from 1.3.2011 and then randomized to the intervention group and the control group in the unit of school using computer generated numbers.

All teachers filled in the first questionnaire and send it back to the investigator in 1 week. 3 copies of the same educational poster were given to the intervention schools, these schools were requested to display them in 1. the medical room 2. staff common room and 3 anywhere that information was usually placed for the teachers. No poster was given to the control group. After 2 weeks, the posters were removed by the teacher in charge. The same questionnaire was filled in by all the teachers in both groups and sent back in 1 week. The data were processed to show whether the poster was effective to improve the knowledge of the teachers. The study was complied with Declaration of Helsinki and ICH GCP guidelines

Primary outcome measures the score of the questionnaire

ELIGIBILITY:
Inclusion Criteria:

* The targeted group of this study included teachers working in primary (US grade1-6) and secondary (US grade 7-12 plus 1 year) schools in Hong Kong, who can read Chinese or English.

Exclusion Criteria:

* cannot read English or Chinese

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
questionnaire score | 2 weeks
  Score - The questionnaire in a related survey - Emergency management of dental trauma: knowledge of Hong Kong primary and secondary school teachers. Young et al. Hong Kong Med J 2012;18:362-70. Chinese and English - 2 sections - 14 questions. - basic demographic information, whether the respondents had received formal first aid training or acquired dental trauma information and whether they thought that they could distinguish deciduous teeth from permanent teeth and management of dental traumatic injuries. The questionnaire was pilot-tested on 81 teachers for length and comprehensibility and was pre-tested before adoption. The face validity was established by expert opinion. The reliability was tested on 41 teachers from a school (14 days), 40 paired questionnaires test-retest reliability, paired t test mean difference between the scores from the 1st and 2nd questionnaires was 0.275. The P value of the t test was 0.4559, The Pearson's product moment correlation coefficient was 0.6887.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Young, BDS MPH, Principal Investigator — The University of Hong Kong
Locations (1):
- Primary and Secondary Schools, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Young C, Wong KY, Cheung LK. Effectiveness of educational poster on knowledge of emergency management of dental trauma-part 1. Cluster randomised controlled trial for primary and secondary school teachers. PLoS One. 2013 Sep 11;8(9):e74833. doi: 10.1371/journal.pone.0074833. eCollection 2013. PMID 24147154